CLINICAL TRIAL: NCT06583018
Title: A Brief and Blended Mindfulness-based Lifestyle Counselling Programme (B-Mindful-Life) for Behavioural Risk Modification Among Caregivers of People With Neurodegenerative Disorders: A Pilot Randomised Controlled Trial
Brief Title: Mindfulness-based Lifestyle Modification Programme for Caregivers of People With Neurodegenerative Disorders: A Pilot Randomised Controlled Trial
Acronym: B-Mindful-Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: health bureau, hong kong (Unknown)
Responsible Party: Principal Investigator, Kwok Yan Yan, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08220157
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Caregiver
Keywords: caregivers; behavioral risk; physical activity; mindfulness; ecological momentary; neurodegenerative diseases; lifestyle
MeSH Terms: conditions — Motor Activity; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief and Blended Mindfulness-based Lifestyle counselling programme (B-Mindful-Life) (Experimental): (i) In-Person Mindfulness-based Group Sessions: Two 3-hour group-based session in week 1 and week 5 focused on experiential mindfulness practices. Participants will enhance their self-awareness of positive, neutral, and negative body sensations, feelings, and thoughts while engaging in healthy behaviors, particularly physical activity.
  (ii) Ecological Momentary Interventions (EMI): Personalized mindfulness-based lifestyle counseling delivered through instant messages, with chat-based support throughout the 8-week intervention period.
  (iii) Activity Monitoring: All participants will wear an accelerometer-based wristband activity tracker to monitor their physical activity in daily life.
- Brief lifestyle education (Active Comparator): (i) In-person Lifestyle Education Session: A 3-hour group-based session in week 1 focused on general education on lifestyle modification.
  (ii) Activity Monitoring: All participants will wear an accelerometer-based wristband activity tracker to monitor their physical activity in daily life.
  Interventions: Behavioral: In-person Lifestyle Education Session; Device: Activity Monitoring

INTERVENTIONS:
Behavioral: In-Person Mindfulness-based Group Sessions — The 3-hour group-based session in week 1 focuses on experiential mindfulness practices, and a booster session in week 5 further consolidates these mindfulness techniques, reinforces mindful, healthy lifestyle, and provides peer support. Participants will enhance their self-awareness of positive, neutral, and negative body sensations, feelings, and thoughts while engaging in healthy behaviors, particularly physical activity.
Behavioral: Ecological Momentary Interventions (EMI) — Participants will receive personalized instant messages with chat-based support throughout the 8-week intervention period. The message content is guided by existing international lifestyle modification guidelines and the Integrated Body-Mind-Spirit Model. The pre-set frequency of regular message delivery is five times per week. The schedule of message delivery will be personalized according to the participants' on-going needs/preferences over the intervention period. Chat-based support will be provided by trained research assistants, who will utilize motivational interviewing techniques to enhance participant compliance and effectiveness.
Behavioral: In-person Lifestyle Education Session — A 3-hour group-based session in week 1 focused on general education on lifestyle modification based on the HEARTS technical package as recommended by the WHO, and will only receive reminder messages for the two assessment follow-ups. No chat-based support will be provided.
  Arms: Brief lifestyle education
Device: Activity Monitoring — All participants will wear an accelerometer-based wristband activity tracker to monitor their physical activity in daily life.
  Arms: Brief lifestyle education

SUMMARY:
Over 80% of caregivers for individuals with neurodegenerative diseases (ND) engage in significant risk behaviors, particularly physical inactivity, which increases the risk of cardiometabolic diseases (CMD) by 30% and reduces life expectancy by 4-8 years. Despite the health benefits of maintaining healthy behaviors, awareness of behavioral risk management among healthcare professionals and the public is low, and research on this topic for ND caregivers is limited. Given that physical activity (PA) is the most prevalent modifiable risk factor, timely intervention is essential.

International guidelines prioritize PA as a key strategy for caregiver health. However, existing PA interventions often struggle with low compliance due to the physical and emotional challenges caregivers face. Our research group actively explores the health-regulating and enhancing effects of integrative mind-body modalities, particularly mindfulness, which may promote and sustain healthy behaviors by improving attentional regulation and psychological flexibility. Mindfulness-based lifestyle modification might help caregivers better manage physical discomfort, stress, and self-limiting beliefs, thereby supporting sustained PA.

The World Health Organization advocates for non-communicable disease (NCD) prevention through brief lifestyle interventions, such as ecological momentary interventions (EMI), which use mobile messaging (e.g., WhatsApp) to deliver personalized health content. This method is particularly valuable for caregivers who find it difficult to access traditional services due to their responsibilities.

This pilot randomized clinical trial aims to evaluate the feasibility and acceptability of an EMI-enhanced "Brief and Blended Mindfulness-based Lifestyle Counselling Programme" (B-Mindful-Life) compared to brief lifestyle education for increasing PA among Chinese ND caregivers. The primary outcome will be the feasibility (rates of recruitment, eligibility, refusal, and retention at 2 and 5 months), and acceptability measures (adherence, incidence of adverse events, and satisfaction with intervention).

ELIGIBILITY:
Inclusion Criteria:

* adults who self-identify as the primary caregivers of ND patients for ≥3 months,
* experience of at least moderate stress as indicated by a PSS score ≥14,
* have a mobile device (e.g., smartphone, tablet, and laptop) with Internet access, and
* able to read and communicate in Chinese and give written consent

Exclusion Criteria:

* a self-reported exercise regimen of great than 150 minutes/week of MVPA (according to the American College of Sports Medicine guidelines),
* have received (within the past 6 months) or are receiving other physical and/or psychosocial interventions,
* pregnancy or within 6 months of postpartum,
* contraindications (e.g., current diagnosis of psychiatric illness according to the DSM IV-TR, DSM-V, or ICD-10) or severe comorbidities (e.g., severe hearing/vision/cognitive impairment) that might limit full participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  Recruitment rate will be calculated as the number of participants who consented to participate in the study divided by the number of eligible participants
Incidence of adverse events | From baseline to the end of the study period at 5 months.
  The incidence of adverse events refers to the occurrence of undesirable experiences or side effects that arise during a clinical trial. It is measured by the number of new adverse events reported during the study period relative to the total number of participants in the study.
  Adverse events are defined as any negative reactions or complications that participants experience, which may be related to the intervention, including but not limited to physical, psychological, or emotional effects.
Retention rate | Baseline, 2 months, and 5 months
  Retention rate will be calculated as the number of participants providing the outcomes of interest divided by the number of randomised participants.
Adherence/ engagement rate | From baseline to the end of intervention at 2 months
  For both groups, the adherence rate will be calculated as the number of participants who attend the group sessions divided by the number of randomized participants.
  For the experimental group, the engagement rate will be calculated as the percentage or frequency of regular messages that are received or replied to by participants using the quick reply button, emojis, or free-text responses. Additionally, it will include the time spent, frequency, and percentage of participants who utilize the chat-based support during the 8-week intervention period.
Satisfaction with intervention | 1-week (the end of the group session), 2-month (the end of the EMI-intervention, for experimental group only)
  Satisfaction will be measured quantitatively by a questionnaire rating on four key domains: usefulness of treatment, opinion of the intervener, perceived improvement and likelihood to recommend the treatment to others, on a 5-point scale. High scores indicating high satisfaction.

SECONDARY OUTCOMES:
Mean change of time spent on 10-minute bout MVPA over a 7-day period | Baseline, 2 months, and 5 months
  For caregivers only, measured by the accelerometer-based wristband activity tracker. The data will be considered valid if the participants wear the activity tracker for ≥10 hours/day for ≥5 days over a 7-day period.
Mean change of time spent on total MVPA over a 7-day period | Baseline, 2 months, 5 months
  For caregivers only, measured by the accelerometer-based wristband activity tracker. The data will be considered valid if the participants wear the activity tracker for ≥10 hours/day for ≥5 days over a 7-day period.
Mean change of time spent on sporadic MVPA over a 7-day period | Baseline, 2 months, 5 months
  For caregivers only, measured by the accelerometer-based wristband activity tracker. The data will be considered valid if the participants wear the activity tracker for ≥10 hours/day for ≥5 days over a 7-day period.
Mean change of average steps per day over a 7-day period | Baseline, 2 month, 5 months
  For caregivers only, measured by the accelerometer-based wristband activity tracker. The data will be considered valid if the participants wear the activity tracker for ≥10 hours/day for ≥5 days over a 7-day period.
Health-related quality of life | Baseline, 2 months, and 5 months
  For both caregivers and care recipients, measured by EuroQol 5-dimension 5-level questionnaire (EQ-5D-5L). The questionnaire comprises two main components: a description of health status across 5 dimensions (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression), and a numeric value representing the overall health status perceived by the respondents (EQ-VAS). Each dimension is rated from 0 (no problems) to 4 (extreme problems). The scores across the 5 dimensions will be transformed into a utility score based on a validated EQ-5D-5L value set for the Chinese population, with a higher utility score indicating a better health state.
  The EQ-VAS records an individual's self-rated health on a numeric analogue visual scale, ranging from 0 (the worst health) to 100 (the best health).
Self-reported level of physical activity | Baseline, 2 months, and 5 months
  For caregivers only, measured by International Physical Activity Questionnaire - Short Form. Continuous scores will be calculated according to the standard scoring protocol, which transforms various physical activities into metabolic equivalent (MET)-minutes/week. A higher MET-minutes/week indicates a higher level of physical activity Based on the duration of different physical activities and the calculated MET-minutes/week, participants can also be classified into three categories: Low, Moderate, and High levels of physical activity.
Percieved stress level | Baseline, 2 months, and 5 months
  For caregivers only, measured by Perceived Stress Scale. Each item is rated on a 0-4 scale (0=never, 4=very often). The total score ranges from 0-40. Higher score indicates higher level of stress. A total score ≥14 indicates moderate level of perceived stress, and a total score ≥27 indicates high level of perceived stress.
Caregiver burden | Baseline, 2 months, and 5 months
  For caregivers only, measured by the 12-item Zarit Burden Interview - Short Version (ZBI-SV). Each item is rated on a 0-4 scale (0=Never, 4=Very Often). The total score ranges from 0-48. Higher score indicates heavier caregiver burden. Three domains of ZBI-SV perceived role strain, self-criticism, and negative emotion will also be assessed.
Anxiety | Baseline, 2 months, and 5 months
  For caregivers only, measured by General Anxiety Disoder - 7 (GAD-7). Each item is rated on a 0-3 scale (0=not at all, 4=nearly every day). The total score ranges from 0-21. Higher score indicates higher level of anxiety. A total score ≥10 indicates possible anxiety.
Depression | Baseline, 2 months, and 5 months
  For caregivers only, measured by Patient Health Questionnaire - 9 (PHQ-9). Each item is rated on a 0-3 scale (0=not at all, 4=nearly every day). The total score ranges from 0-27. Higher score indicates higher level of depression. A total score ≥10 indicates possible major depression.
Mindfulness | Baseline, 2 months, and 5 months
  For caregivers only, measured by 20-item Five-facet Mindfulness Questionnaire - Short Form (FFMQ-SF). Each item is rated on 1-5 scale (1=Never, 5=Very Often). The total score ranges from 20-100. Higher score indicates higher level of trait mindfulness. In addition, five domains of the FFMQ-SF, namely observing, describing, acting with awareness, non-judgment of inner experience, and non-reaction to inner experience will be assessed.
Self-care behaviors | Baseline, 2 months, and 5 months
  For caregivers only, measured by 20-item Self-Care Inventory (SCI). Each item is rated on a 1 to 5 scale (1=Never, 5=Always). 3 domains of the SCI, namely self-care maintenance, self-care monitoring, and self-care management will be assessed. The score of each domain is derived from the raw summative score using the scoring algorithm proposed by the scale developer, which ranges from 0 to 100. A higher score on the SCI indicates better engagement in self-care in the corresponding domain.
Self-care efficacy | Baseline, 2 months, and 5 months
  For caregivers only, measured by the 10-item Self-Care Self-Efficacy Scale (SCSES). Each item is rated on a 1 to 5 scale (1=No Confident, 5=Extremely Confident). The total score ranges from 10-50. Higher score in SCSES indicates higher level of self-care efficacy.
Attention and meditation levels | Baseline, 2 months, and 5 months
  For caregivers only, measured using a validated electroencephalogram-based headband tracker. Participants will wear the headband with assistance from the outcome assessor before following a standardized audio-guided protocol. Attention and meditation levels will be assessed using a 0-100 rating scale, where a higher score indicates increased focused attention and meditation status, respectively.
Support care needs | Baseline, 2 months, and 5 months
  For care recipients only, meausred by the 10-item Palliative care Outcome Scale (POS). The 10 items assess physical symptoms, emotional, psychosocial and spiritual needs, provision of information and practical concerns. Each item is rated on a 0 - 4 scale (0=No burden, 4=Overwhelming problems). The total score ranges from 0-40. Higher score indicates greater unmet support care needs.

OTHER OUTCOMES:
Participant expereince and perception of the intervention | Within three months after the end of the intervention
  For the experimental group participants, a semi-structured individual interview will be conducted to explore their perceptions and experiences of the intervention. The focus will be on understanding the perceived effects, how and why the intervention works or does not work, and the conditions that may influence their motivation, acceptability, and real-life application.

CONTACTS AND LOCATIONS:
Overall Officials: Jojo Yan Yan Kwok, BNurs, MPH, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, LKS Faculty of Medicine, The University of Hong Kong, Pokfulam, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data supporting the findings of this study are available upon request from the principal investigator, Dr. Kwok. These data are not publicly available, as they contain information that could compromise the privacy of research participants.